CLINICAL TRIAL: NCT04598685
Title: Early Vascular Ageing in the YOUth - An Observational Study Into the Predictors of Atherosclerotic Changes in Adolescents
Brief Title: Early Vascular Ageing in the YOUth
Acronym: EVA4YOU
Status: Completed | Type: Observational
Sponsor: VASCage GmbH (Other)
Collaborators: Medical University Innsbruck (Other); Tirol Kiniken GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: EVA4YOU
Record Dates: First submitted 2020-09-23; First posted 2020-10-22 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Atherosclerosis; Cardiovascular Risk Factor; Cardiovascular Diseases; Cardiovascular Pathology; Life Style; Vascular Diseases; Vascular Stiffness; Non-Alcoholic Fatty Liver Disease; Hypertension; Obesity; Overweight; Headache; Sleep; Sleep Disorder
Keywords: Cardiovascular Diseases; Cardiovascular Risk Factor; Atherosclerosis; Cardiovascular Pathology; Life Style; Vascular Diseases; Early Vascular Ageing; Vascular Stiffness; Intima-Media Thickness; Non-Alcoholic Fatty Liver Disease; Ultrasonography; Liver Elastography; Bioimpedance; Blood Pressure; Body Mass Index; Headache; Sleep; Adolescence
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Vascular Diseases; Non-alcoholic Fatty Liver Disease; Hypertension; Obesity; Overweight; Headache; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — * Blood: (lipidome, proteome)
    * whole blood (DNA)
    * Serum
    * Plasma
  * Stool (gut microbiome)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single-center observational study on adolescents to determine predictors of the early steps of the formation of atherosclerosis and to quantify their influence on Intima-Media-Thickness of the carotid artery and the aorta and on the Pulse-Wave Velocity.

A long-term follow-up by means of record linkage is furthermore planned to evaluate the effect of early atherosclerosis and the cardiovascular risk profile on future morbidity with a special focus cardio- and cerebrovascular events.

DETAILED DESCRIPTION:
EVA4YOU is a cross-sectional study enrolling 3000 students and apprentices aged between 14 and 19 years. Examinations are conducted at schools and companies throughout Tyrol, Austria and include laboratory measurements; standardized medical interviews; anthropometry; liver elastography; ultrasonography of the carotid artery and the aorta, and blood pressure, bioelectrical impedance; visceral abdominal fat-tissue-thickness measurement, pulse-wave velocity measurements.

The study hypothesis is that the cardiovascular risk factors measured already influence the formation of atherosclerosis (measured as carotid and aortic Intima-Media Thickness and Pulse-Wave-Velocity) in adolescents.

A long-term follow-up by means of record linkage is furthermore planned to evaluate the effect of early atherosclerosis and the cardiovascular risk profile on future morbidity with a special focus cardio- and cerebrovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents at the age of 14 to 19 years
* Signed informed consent of subjects (and legal guardian if subject < 18 years of age)

Exclusion Criteria:

* Persons, who are suspended upon a court order or upon other legal processes or are accommodated according to the Hospitalization Act, or for whom a custodian is appointed (or appointment is initiated).
* Persons with impaired power of judgment
* Persons who are currently engaged in military or community service

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: students and apprentices aged 14-19 years
Sampling Method: Non-Probability Sample
Enrollment: 1517 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Determinants of Intima-Media Thickness (carotid and aortic) | Day 1
  Predictors to be examined include: Blood Pressure, BMI/body composition, Smoking, Physical Activity, Family History, Lipid and Glucose Metabolism, NAFLD, Diet, Sex, Age used as predictors in multiple regression analysis
Determinants of the Pulse-Wave Velocity [m/s] | Day 1
  Predictors to be examined include: Blood Pressure, BMI/body composition, Smoking, Physical Activity, Family History, Lipid and Glucose Metabolism, NAFLD, Diet, Sex, Age used as predictors in multiple regression analysis
  The pulse-wave velocity [m/s] is measured by using the Vicorder, an oscillometric pulse-wave measurement device.

SECONDARY OUTCOMES:
Predictors of later cardio- and cerebrovascular disease (events and mortality) by record linkage | every 2-5 years, on average for the duration of 50 years
  Occurence of major adverse cardiovascular events (yes/no, time to event), assessed by means of automated detection of these events by record linkage
Prevalence of traditional cardiovascular risk and lifestyle factors and descripition of high-risk populations | Day 1
Time trends in risk profiles by comparison to data from the Early Vascular Ageing (EVA) study, NCT03929692 | 8 years

OTHER OUTCOMES:
The effect of primary headache disorders on Intima-Media Thickness [µm] | Day 1
  Primary Headache Disorders are assessed by means of structured medical questionnaires in a physician-guided interview and classified according to the ICHD-3 Classification System. Differences in terms of vessel wall thickness [µm], measured ultrasonographically, are compared across the different primary headache diagnoses.
The effect of primary headache disorders on Pulse-Wave Velocity [m/s] | Day 1
  Primary Headache Disorders are assessed by means of structured medical questionnaires in a physician-guided interview and classified according to the ICHD-3 Classification System. Differences in terms of pulse-wave velocity [m/s], measured with use of an oscillometric pulse-wave measurement device, are compared across the different primary headache diagnoses.
The effect of the gut microbiome on the cardiovascular risk profile. | Day 1
  Structure and composition of the Microbiom using 16S metagenomics and shotgun metagenomics and are evaluate for their interrelationship with cardiovascular risk parameters (such as hypertension, smoking, dyslipidemia, impaired glucose tolerance, overweight/obesity, sedentary lifestyle, unhealthy dietary habits, ...).
  Where appropriate additional functional insight will be obtained by metabolomics (gas chromatography and MR chromatography).
The effect of the gut microbiome on Intima-Media Thickness [µm] | Day 1
  Structure and composition of the Microbiom using 16S metagenomics and shotgun metagenomics and are assessed using stool samples and are evaluate for their influence on intima-media thickness, measured via ultrasonography. Where appropriate additional functional insight will be obtained by metabolomics (gas chromatography and MR chromatography).
The effect of prenatal and infant development (early life risk factors) on Intima-Media Thickness [µm]. | Day 1
  Prenatal and infant development is assessed using records from mother-child-booklets and a questionnaire for the mother and the influence on intima-media thickness, measured using ultrasonography, is evaluated.
The effect of prenatal and infant development (early life risk factors) on the cardiovascular risk profile. | Day 1
  Prenatal and infant development is assessed using records from mother-child-booklets and a questionnaire for the mother and the influence on the cardiovascular risk profile (i.e. existence of cardiovascular risk factors such as hypertension, smoking, dyslipidemia, impaired glucose tolerance, overweight/obesity, sedentary lifestyle, unhealthy dietary habits, ...) is evaluated.
Prevalence of headache disorders (especially primary headache disorders) in adolescents | Day 1
  Headache Disorders are assessed by means of structured medical questionnaires (including duration, frequency, intensity, headache characteristics and concomitant symptoms) in a physician-guided interview and classified according to the ICHD-3 Classification System.
Risk factors for primary headache disorders in adolescents | Day 1
  Headache Disorders are assessed by means of structured medical questionnaires (including duration, frequency, intensity, headache characteristics and concomitant symptoms) in a physician-guided interview and classified according to the ICHD-3 Classification System.
  Risk factors to be assessed for their association with primary headache disorders include: Alcohol, caffeine and nicotine consumption, physical activity, obesity, dysfunctional familial situation, mental comorbidities are assessed in structured physician-guided interviews and questionnaires.
Risk factors for the chronification of primary headache-disorders | Day 1
  Headache Disorders are assessed by means of structured medical questionnaires (including duration, frequency, intensity, headache characteristics and concomitant symptoms) in a physician-guided interview and classified according to the ICHD-3 Classification System.
  Risk factors to be assessed for their effect on chronification of primary headache disorders include: Alcohol, caffeine and nicotine consumption, physical activity, obesity, dysfunctional familial situation, mental comorbidities are assessed in structured physician-guided interviews and questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Knoflach, MD, Principal Investigator — Medical University Innsbruck
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data can be shared in academic cooperations. Request for data can be addressed to the principal investigators with an appropriate research question.

REFERENCES:
- [Derived] Messner A, Nairz J, Kiechl SJ, Winder B, Hochmayr C, Granna J, Egger A, Griesmacher A, Geiger R, Knoflach M, Kiechl-Kohlendorfer U; Early Vascular Ageing in the YOUth (EVA4YOU) Study Group. Thresholds of fat mass index percentiles and their association with cardiovascular risk in adolescents: Results from the EVA4YOU study. Nutr Metab Cardiovasc Dis. 2026 Feb;36(2):104408. doi: 10.1016/j.numecd.2025.104408. Epub 2025 Oct 8. PMID 41087203
- [Derived] Messner A, Nairz J, Kiechl S, Winder B, Pechlaner R, Geiger R, Knoflach M, Kiechl-Kohlendorfer U; EVA4YOU Tyrol Study Group. Comparison of body mass index and fat mass index to classify body composition in adolescents-The EVA4YOU study. Eur J Pediatr. 2024 May;183(5):2203-2214. doi: 10.1007/s00431-024-05474-x. Epub 2024 Feb 22. PMID 38386029